CLINICAL TRIAL: NCT00797381
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety, Tolerability of MK-0518 in Treatment-Experienced HIV-1 Infected Adult Patients With Hemophilia
Brief Title: Efficacy and Safety of MK-0518 in Treatment-Experienced HIV-1 Infected Adult Patients With Hemophilia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Public Health Clinical Center (Other Government)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Shanghai Public Health Clinical Center, Shanghai Public Health Clinical Center
Other Study IDs: CN2009
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Last update posted 2008-11-25 (Estimated); Status verified 2008-11

CONDITIONS: HIV Infection; Hemophilia A
Keywords: MK-0518; HIV; AIDS; hemophilia; treatment experienced
MeSH Terms: conditions — HIV Infections; Hemophilia A; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 3 ml plasm of each subject on week 4,8,12 and 24
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1
- 2

SUMMARY:
This is an randomized, double-blind, placebo-controlled study to assess the safety, tolerability and efficacy of MK-0518 compared to placebo when combined with other antiretroviral drugs, in treatment-experienced HIV-infected patients with hemophilia.

Subjects enrolled in the study sign the consent form, then are randomly assigned to MK-0518 400 mg twice daily plus optimized background therapy (OBT) group or placebo plus OBT group.Each group concludes at least 50 subjects. For each patient, detection of HIV viral load and CD4+ T lymphocyte count is done at screening, and at weeks 4, 8, 12 and 24. The safety profile of MK-0518 is monitored according to patients' complaints and the results of physical and laboratory examinations.

The safety and efficacy of MK-0518 400 mg b.i.d. compared to placebo, both in combination with OBT, will be assessed by review of the accumulated study data in HIV-infected patients with hemophilia.

DETAILED DESCRIPTION:
1. Objective

   To assess the safety, tolerability and efficacy of MK-0518 compared to placebo when combined with other antiretroviral drugs, in treatment-experienced HIV-infected patients with hemophilia.
2. Background and Significance

Current anti-HIV drugs are mainly reverse transcriptase inhibitors, which include nucleoside reverse transcriptase inhibitors(NRTIs) and non-nucleoside reverse transcriptase inhibitors(NNRTIs), and protease inhibitors(PIs). However, HIV can become rapidly resistant to them due to its high rate of mutation while replicating, which forces people to seek new targets for anti-HIV therapy continually. Integrase is an another enzyme essential for HIV reproduction. To inhibit integrase activity is an effective measure to suppress HIV replication. MK-0518(Raltegravir）was approved by the United States Food and Drug Administration(FDA) on October 12th 2007 due to its potent antiviral activity and became the first-to-market integrase inhibitor.Compared with other antiviral drugs, it has new action mechanism and target site, so there is no cross resistance between it and them, which makes it a good option for patients with multi-drug resistant HIV strains. HIV infection is very common in hemophiliac patients who need continuous infusion of clotting products,and the chance of getting HIV infection for hemophilia patients is very high, especially before 1985 when non-virus-inactivated factor concentrates were widely used. Many hemophilia patients were infected with HIV, and AIDS became their main cause of death.The recommended first-line antiretroviral regimen for HIV/AIDS patients with hemophilia concludes two NRTIs and one NNRTIs, while protease inhibitors are not recommended to use in these patients, because they are likely to worsen bleeding tendency. So, if HIV/AIDS patients with hemophilia are resistant to NRTIs and NNRTIs, there are few remaining options for them to choose as part of second-line drugs. However, MK-0518，a drug with novel anti-HIV mechanism different with NRTIs and NNRTIs, may be used in HIV/AIDS patients with hemophilia as the second-line drug.

3． Study design

1. Patients Enrollment
2. Patients enrolled in the study sign consent form
3. Select an optimized background therapy(OBT) for each subject
4. Randomization: patients are randomly assigned to MK-0518 400 mg twice daily plus OBT group or placebo plus OBT group, each group concludes at least 50 subjects.
5. Data collection: for each patient, detection of HIV viral load and CD4+ T lymphocyte count is done at screening, and at weeks4, 8, 12, 16, and 24. The safety profile of MK-0518 is monitored according to patients' complaints and the results of physical and laboratory examinations.
6. Endpoints of study: The primary endpoint is the the safety and tolerability of MK-0518 400 mg b.i.d. compared to placebo, both in combination with OBT.The secondary endpoint is antiretroviral activity of MK-0518 400 mg b.i.d. compared to placebo, both in combination with OBT.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected patients with hemophilia aged over 18 who have failed previous antiretroviral treatment are eligible.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: treatment-experienced HIV-1 infected adult patients with hemophilia
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-05; Primary Completion 2010-10 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
The safety and tolerability of MK-0518 400 mg b.i.d. compared to placebo, both in combination with OBT, assessed by review of the accumulated safety data in HIV-infected patients with hemophilia. | 24 weeks

SECONDARY OUTCOMES:
Antiretroviral activity of MK-0518 400 mg b.i.d. compared to placebo, both in combination with OBT. | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hongzhou Lu, PhD, Principal Investigator — Shanghai Public Health Clinical Center
Locations (1):
- Shanghai Public Health Clinical Center, Shanghai, Jinshan, China